CLINICAL TRIAL: NCT03646812
Title: Glycemic and Insulinemic Response of Pasta Products in Comparison to Asian
Brief Title: Glycemic and Insulinemic Response of Pasta Products in Comparison to Asian Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Barilla Singapore Pte Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018/00622
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Glucose Reference 1 (Other): 50g of glucose dissolved in 250ml of water to be consumed.
  Interventions: Other: Glucose Reference 1
- Glucose Reference 2 (Other): 50g of glucose dissolved in 250ml of water to be consumed.
  Interventions: Other: Glucose Reference 2
- Glucose Reference 3 (Other): 50g of glucose dissolved in 250ml of water to be consumed.
  Interventions: Other: Glucose Reference 3
- Semolina Penne (Experimental): 70g of semolina penne boiled in 1 Litre of water for 11 minutes. Drained and consume immediately.
  Interventions: Other: Semolina Penne
- Wholegrain Penne (Experimental): 76g of wholegrain penne boiled in 1 Litre of water for 9 minutes. Drained and consume immediately.
  Interventions: Other: Wholegrain Penne
- Semolina Spaghetti (Experimental): 71g of semolina spaghetti boiled in 1 Litre of water for 8 minutes. Drained and consume immediately.
  Interventions: Other: Semolina Spaghetti
- Wholegrain Spaghetti (Experimental): 76g of wholegrain spaghetti boiled in 1 Litre of water for 8 minutes. Drained and consume immediately.
  Interventions: Other: Wholegrain Spaghetti
- Jasmine rice (Experimental): 63g of rice cook with 150g of water. Served and consume immediately.
  Interventions: Other: Jasmine Rice
- Asian Noodles (Experimental): 92.4g of Asian Noodles cook in boiling water for 45 seconds. Drained and consume immediately
  Interventions: Other: Asian Noodles

INTERVENTIONS:
Other: Glucose Reference 1 — Glucose contains 50g of available carbohydrates
  Arms: Glucose Reference 1
Other: Glucose Reference 2 — Glucose contains 50g of available carbohydrates
  Arms: Glucose Reference 2
Other: Glucose Reference 3 — Glucose contains 50g of available carbohydrates
  Arms: Glucose Reference 3
Other: Semolina Penne — Semolina Penne contains 50g of available carbohydrates
  Arms: Semolina Penne
Other: Wholegrain Penne — Wholegrain Penne contains 50g of available carbohydrates
  Arms: Wholegrain Penne
Other: Semolina Spaghetti — Semolina Spaghetti contains 50g of available carbohydrates
  Arms: Semolina Spaghetti
Other: Wholegrain Spaghetti — Wholegrain Spaghetti contains 50g of available carbohydrates
  Arms: Wholegrain Spaghetti
Other: Jasmine Rice — Jasmine Rice contains 50g of available carbohydrates
  Arms: Jasmine rice
Other: Asian Noodles — Asian Noodles contains 50g of available carbohydrates
  Arms: Asian Noodles

SUMMARY:
The aim of the study is to determine the glycaemic and insulinaemic index of pasta products and local foods. It is hypothesized that different pasta cuts and wholegrain composition of pasta and local foods have different GI depending on the nature of the carbohydrate content and the food structure within each food.

DETAILED DESCRIPTION:
There will be a total of 9 test sessions and each session will last up to 3.5 hours. The order of sessions will be determined with an online randomizer. At each test session, the following procedures will be performed: two finger-prick blood samples, five minutes apart to measure baseline blood glucose and insulin concentrations Subject will be served the test food and to consume within15 minutes Following the test meal, blood samples will be collected at the following time points: 15, 30, 45, 60, 90, 120, 150 and 180min for glucose measurements and insulin measurements will be collected at 30, 60, 90, 120, 150 and 180min.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Asian - Indian and Chinese ethnicity
* Age between 21-40 years
* Body mass index between 18.5 to 25 kg/m2
* Normal blood pressure (<140/90 mmHg)
* Fasting blood glucose < 6 mmol/L

Exclusion Criteria:

* Is a current smoker
* Is currently pregnant
* Have any metabolic diseases (such as diabetes, hypertension etc)
* Have known glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Have medical conditions and/or taking medications known to affect glycemia(glucocorticoids, thyroid hormones, thiazide diuretics)
* Have any major organ dysfunction (e.g. cardiovascular, respiratory, hepatic, renal, gastrointestinal) that may influence taste, olfaction, appetite, digestion, metabolism, absorption or elimination of test foods, nutraceutical or drug
* Have any severe food allergy (e.g. anaphylaxis to peanuts)
* Have any known allergies to any food components of the study protocol
* Have active Tuberculosis (TB) or currently receiving treatment for TB
* Have any known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Is a study team member or an immediate family of any study team member. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* enrolled in a concurrent research study judged not to be scientifically or medically compatible with the study.
* Have partake in sports at the competitive and/or endurance levels
* Have intentionally restrict food intake

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Glucose | up to 180 minutes
  Blood will be collected and measured using hemocue analyzer.
Insulin | up to 180 minutes
  Blood will be collected and measured using COBAS analyzer.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No